CLINICAL TRIAL: NCT02452268
Title: A Phase 1 Study of Subcutaneous Recombinant Human NIZ985 ((hetIL-15) (IL15/sIL-15Ra)) Alone and in Combination With PDR001 in Adults With Metastatic Cancers
Brief Title: A Phase I/Ib Study of NIZ985 in Combination With PDR001 in Adults With Metastatic Cancers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: business decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNIZ985X2102J; NIZ985X2102J (Other: Novartis)
Record Dates: First submitted 2015-03-02; First posted 2015-05-22 (Estimated); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Metastatic and Advanced Solid Tumors
MeSH Terms: conditions — Neoplasm Metastasis | interventions — spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NIZ985 (Experimental): * Single treatment arm, dose escalation administered subcutaneously (SC) on MWF for 2 consecutive weeks.
  * Cycle length 28 days.
  * Occurrence of a dose-limiting toxicity (DLT) leads to the expansion to 6 subjects.
  * MTD is the dose prior to the dose level where ≥ 2/6 subjects have a DLT.
  * Following identification of the MTD / RDE, dose expansion will follow.
  Interventions: Drug: NIZ985
- NIZ985 + PDR001 (Experimental): * The phase Ib dose escalation portion of the study will consist of a fixed dose (400 mg, IV infusion, Q4W) of PDR001 and escalating doses of NIZ985 (hetIL-15) to evaluate safety, tolerability and determine the MTD and/or RDE of the combination to be used in expansion cohorts.
  * On days when PDR001 and NIZ985 are administered on the same day, PDR001 will be administered first. NIZ985 will be administered after the PDR001 infusion has been completed.
  * Information on the preparation and administration of PDR001 is found in the PDR001 pharmacy manual.
  Interventions: Drug: PDR001

INTERVENTIONS:
Drug: NIZ985 — Subcutaneous administration of hetIL-15 three times a week for two consecutive weeks
  Other Names: IL-15/sIL-15Ra, heterodimeric IL-15
  Arms: NIZ985
Drug: PDR001 — • PDR001 is a human monoclonal antibody (MAb) administered day 1 of each cycle
  Arms: NIZ985 + PDR001

SUMMARY:
Phase I/Ib multicenter clinical trial. Single agent dose escalation of NIZ985 followed by expansion. Second escalation of NIZ985 in combination with PDR001 followed by expansion

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed solid tumor malignancy that is metastatic or unresectable and have progressed on at least 1 prior therapy and for whom standard curative or palliative measures do not exist or are associated with minimal subject survival benefit.

   Evaluable or measurable disease, defined as by Response Evaluation Criteria in Solid Tumors (RECIST).
2. Recovered to ≤ grade 1 NCI CTCAE version 4.0 from toxicity of prior chemotherapy or biologic therapy administered more than 4 weeks earlier.
3. Subjects on bisphosphonates for any cancer or on hormone therapy for prostate cancer may continue this therapy. However, subjects with prostate cancer must have confirmed metastatic disease that has progressed despite hormonal therapy producing castrate levels of testosterone.
4. Age ≥18 years.
5. ECOG performance status ≤1 (Karnofsky ≥70%).
6. Normal organ and marrow function:

   * leukocytes ≥3,000/mcL
   * absolute neutrophil count (ANC) ≥1,500/mcL
   * platelets ≥100,000/mcL
   * total bilirubin within normal institutional limits
   * AST/ALT ≤2.5 × ULN
   * creatinine <1.5 × institutional ULN OR
   * creatinine clearance ≥60 mL/min/1.73 m2 for subjects with serum creatinine levels >1.5 × higher than ULN.
7. DLCO/VA and FEV1 ≥ 50% of predicted on PFTs.
8. Subjects with inactive central nervous system (CNS) metastasis are eligible..
9. Women of child-bearing potential and men must agree to use adequate contraception prior to study entry, during the treatment portion of the study and for 4 months after completion of hetIL-15 administration.
10. Able to provide written informed consent.
11. Life expectancy > 3 months.

Exclusion Criteria:

1. Prior IL-15 treatment or cytotoxic therapy, immunotherapy, radiotherapy, major surgery, antitumor vaccines or monoclonal antibodies in the 4 weeks prior or for checkpoint inhibitors such as anti-CTLA-4 or anti PD1/PD-L1 or nitrosoureas or mitomycin C for 6 weeks prior to C1D1.
2. Primary brain cancers or active CNS metastases should be excluded from this clinical trial
3. History of allergic reactions attributed to compounds of similar chemical or biologic composition to hetIL-15.
4. Concurrent anticancer therapy (including other investigational agents) with the exception of hormone therapy for prostate cancer.
5. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, cognitive impairment, active substance abuse, or psychiatric illness/social situations that, in the view of the Investigator, would preclude safe treatment or the ability to give informed consent and limit compliance with study requirements.
6. HIV positive patients.
7. Positive hepatitis B or C serology.
8. History of severe asthma or absolute requirement for chronic inhaled corticosteroid medications.
9. History of autoimmune disease, with the exception of an autoimmune event associated with prior ipilimumab (anti-CTLA-4) therapy that has been completely resolved for more than 4 weeks prior to C1D1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2022-03-07 (Actual)

PRIMARY OUTCOMES:
Assess the dose-limiting toxicity of the single agent NIZ985 and the combination of PDR001 | 28 days

SECONDARY OUTCOMES:
Determine the maximum tolerated dose (MTD) of hetIL-15 as determined by DLTs during Cycle 1. | 28 days
Determine the pharmacokinetic (PK) profile of hetIL-15, including T½ | 28 days
Determine the pharmacokinetic (PK) profile of hetIL-15, including Cmax. | 28 Days
Determine the preliminary anti-tumor activity of hetIL-15 | 8 weeks
  Best overall response (BOR) per RECIST and irRC

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- United States (7):
  - National Cancer Institute National Cancer Institute, Bethesda, Maryland
  - Washington University School of Medicine SC, St Louis, Missouri
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Providence Portland Medical Center SC, Portland, Oregon
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leidner R, Conlon K, McNeel DG, Wang-Gillam A, Gupta S, Wesolowski R, Chaudhari M, Hassounah N, Lee JB, Ho Lee L, O'Keeffe JA, Lewis N, Pavlakis GN, Thompson JA. First-in-human phase I/Ib study of NIZ985, a recombinant heterodimer of IL-15 and IL-15Ralpha, as a single agent and in combination with spartalizumab in patients with advanced and metastatic solid tumors. J Immunother Cancer. 2023 Oct;11(10):e007725. doi: 10.1136/jitc-2023-007725. PMID 37907221
- [Derived] Conlon K, Watson DC, Waldmann TA, Valentin A, Bergamaschi C, Felber BK, Peer CJ, Figg WD, Potter EL, Roederer M, McNeel DG, Thompson JA, Gupta S, Leidner R, Wang-Gillam A, Parikh NS, Long D, Kurtulus S, Ho Lee L, Chowdhury NR, Bender F, Pavlakis GN. Phase I study of single agent NIZ985, a recombinant heterodimeric IL-15 agonist, in adult patients with metastatic or unresectable solid tumors. J Immunother Cancer. 2021 Nov;9(11):e003388. doi: 10.1136/jitc-2021-003388. PMID 34799399
- [Derived] Watson DC, Moysi E, Valentin A, Bergamaschi C, Devasundaram S, Fortis SP, Bear J, Chertova E, Bess J Jr, Sowder R, Venzon DJ, Deleage C, Estes JD, Lifson JD, Petrovas C, Felber BK, Pavlakis GN. Treatment with native heterodimeric IL-15 increases cytotoxic lymphocytes and reduces SHIV RNA in lymph nodes. PLoS Pathog. 2018 Feb 23;14(2):e1006902. doi: 10.1371/journal.ppat.1006902. eCollection 2018 Feb. PMID 29474450
- See also: Study Results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18021